CLINICAL TRIAL: NCT01869582
Title: Safer Births - New Knowledge and Innovations to Decrease Perinatal Mortality and Morbidity Worldwide
Brief Title: Safer Births - Reducing Perinatal Mortality
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Helse Stavanger HF (Other Government)
Collaborators: Muhimbili National Hospital, Tanzania (Unknown); Haydom Lutheran Hospital (Other); Stavanger Acute medicine Foundation for Education and Research, Norway (Unknown); Weill Cornell Medical Collage, USA (Unknown); Laerdal Global Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: Safer Births
Record Dates: First submitted 2013-05-24; First posted 2013-06-05 (Estimated); Last update posted 2020-05-12 (Actual); Status verified 2017-05

CONDITIONS: Fetal Heart Rate Abnormalities; Respiratory Depression; Birth Asphyxia; Neonatal Resuscitation
Keywords: Fetal hypoxia; Birth asphyxia; Neonatal resuscitation
MeSH Terms: conditions — Respiratory Insufficiency; Asphyxia Neonatorum; Fetal Hypoxia | interventions — Fetoscopes; Resuscitation; Echocardiography, Doppler

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Doppler, Fetal heart rate (Experimental): Eligible women in labour randomized to intermittent fetal heart rate assessments using a wind-up, hand-held Doppler
  Interventions: Device: Doppler, Fetal heart rate
- Fetoscope, Fetal heart rate (Experimental): Eligible women in labour randomized to intermittent fetal heart rate assessments using a Pinard fetoscope, which is the current standard management
  Interventions: Device: Fetoscope, Fetal heart rate
- Upright Resuscitator, Resuscitation (Experimental): Non-breathing newborn infants in need of positive pressure ventilation randomized to an Upright Resuscitator
  Interventions: Device: Upright Resuscitator, Resuscitation
- Standard Resuscitator, Resuscitation (Experimental): Non-breathing newborn infants in need of positive pressure ventilation randomized to a standard horizontal Resuscitator, which is the current standard management
  Interventions: Device: Standard Resuscitator, Resuscitation

INTERVENTIONS:
Device: Fetoscope, Fetal heart rate
  Other Names: Pinard fetoscope
  Arms: Fetoscope, Fetal heart rate
Device: Upright Resuscitator, Resuscitation
  Other Names: Laerdal Upright Resuscitator
  Arms: Upright Resuscitator, Resuscitation
Device: Doppler, Fetal heart rate
  Other Names: FreePlay Doppler Ultrasound
  Arms: Doppler, Fetal heart rate
Device: Standard Resuscitator, Resuscitation
  Other Names: Laerdal Neonatal Resuscitator
  Arms: Standard Resuscitator, Resuscitation

SUMMARY:
Safer Births is a research and development collaboration to establish new knowledge and new innovative products to better equip and increase competence of health workers for safer births and increased newborn survival worldwide.

The main objectives are:

To randomize different devices for fetal heart rate assessments. To assess if a novel Newborn Resuscitation Monitor will facilitate newborn resuscitation in a low-resource setting. To determine bag mask ventilation treatment and devices beneficial for neonatal outcome.

ELIGIBILITY:
Inclusion Criteria:

* Randomizing fetal heart rate assessment: Singleton delivery, Term gestation age, Cephalic presentation, Fetal heart rate normal, Cervical dilatation ≤7cm, Consent to participate
* Randomizing bag mask ventilation: infants in need of positive pressure ventilation, Consent to participate

Exclusion Criteria:

* Randomizing fetal heart rate assessment: Placenta abruption/praevia, Ruptured uterus, Morbid Obesity

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20000 (Estimated)
Dates: Start 2013-03 (Actual); Primary Completion 2018-04 (Actual); Study Completion 2018-04 (Actual)

PRIMARY OUTCOMES:
Perinatal Mortality | From start of labour to 7 days postpartum
  Death during or shortly following birth

CONTACTS AND LOCATIONS:
Overall Officials: Hege L Ersdal, MD, PhD, Principal Investigator — Helse Stavanger HF; Hussein L Kidanto, MD, PhD, Principal Investigator — Muhimbili National Hospital; Estomih R Mduma, Manager, Principal Investigator — Haydom Lutheran Hospital
Locations (2):
- Tanzania (2):
  - Haydom Lutheran Hospital, Research Institute, Haydom, Manyara Region
  - Muhimbili National Hospital, Dar es Salaam

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mdoe PF, Ersdal HL, Mduma ER, Perlman JM, Moshiro R, Wangwe PT, Kidanto H. Intermittent fetal heart rate monitoring using a fetoscope or hand held Doppler in rural Tanzania: a randomized controlled trial. BMC Pregnancy Childbirth. 2018 May 4;18(1):134. doi: 10.1186/s12884-018-1746-9. PMID 29728142
- [Derived] Thallinger M, Ersdal HL, Francis F, Yeconia A, Mduma E, Kidanto H, Linde JE, Eilevstjonn J, Gunnes N, Stordal K. Born not breathing: A randomised trial comparing two self-inflating bag-masks during newborn resuscitation in Tanzania. Resuscitation. 2017 Jul;116:66-72. doi: 10.1016/j.resuscitation.2017.04.012. Epub 2017 Apr 17. PMID 28427883